CLINICAL TRIAL: NCT04581395
Title: The Effect of Precurarization With Rocuronium on the Incidence and Severity of Succinylcholine-Induced Fasciculations and Myalgias in a High Volume ERCP Center
Brief Title: The Effect of Pretreatment With Roc on Succinylcholine Myalgias
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Leighan S. Bye, MD, PhD, Assistant Professor of clinical Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1912284619
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Myalgia
Keywords: Myalgias; Fasciculations; succinylcholine; rocuronium; pretreatment; precurarization
MeSH Terms: conditions — Myalgia; Fasciculation | interventions — Control Groups; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization will be performed using Research Randomizer in blocks of 30. The primary investigator will inform the person doing the case as to what group the participants are randomized. Both the participants and the research staff doing assessments will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Not pretreated (Other): Succinylcholine administration with no Rocuronium pre-treatment
  Interventions: Other: non-pretreated Succinylcholine
- Pre-treated 1 minute before succinylcholine administration (Active Comparator): Succinylcholine administration 1 minute following Rocuronium pre-treatment
  Interventions: Drug: succinylcholine 1 minute after rocuronium pretreatment
- Pre-treated 2 minutes before succinylcholine administratjion (Active Comparator): Succinylcholine administratjion 2 minutes following Rocuronium pre-treatment
  Interventions: Drug: succinylcholine 2 minutes following rocuronium pretreatment

INTERVENTIONS:
Other: non-pretreated Succinylcholine — no pretreatment
  Other Names: Control group
  Arms: Not pretreated
Drug: succinylcholine 1 minute after rocuronium pretreatment — 0.05 mg/kg up to 5 mg of rocuronium pretreatment followed by 1.0 mg/kg succinlycholine t = 1 min +/- 10 sec after pretreatment
  Other Names: rocuronium pretreatment 1 minute before succinylcholine administration
  Arms: Pre-treated 1 minute before succinylcholine administration
Drug: succinylcholine 2 minutes following rocuronium pretreatment — 0.05 mg/kg up to 5 mg of rocuronium pretreatment followed by 1.0 mg/kg succinlycholine t = 2 min +/- 10 sec after pretreatment.
  Other Names: rocuronium pretreatment 2 minutes before succinylcholine administration
  Arms: Pre-treated 2 minutes before succinylcholine administratjion

SUMMARY:
Succinylcholine is a medication (depolarizing muscle relaxant) that is used as part of an anesthetic (going to sleep for surgery). This medication can cause significant muscle soreness. Rocuronium is a medication (non-depolarizing muscle relaxant) that some anesthesia providers believe may reduce muscle soreness caused by succinylcholine if given prior, but this has been controversial. Some anesthesiologists pretreat patients with rocuronium before giving patients succinylcholine, and some do not. The purpose of this study is to examine the effect of pretreatment with rocuronium on muscle soreness associated with succinylcholine administration.

DETAILED DESCRIPTION:
After IRB approval from Indiana University Hospital and with written and verbal informed consent from each patient, 300 ASA I, II and III outpatients scheduled for elective Endoscopic Retrograde Cholangiopancreatography (ERCP) under general anesthesia will be enrolled in this randomized-controlled study. The participants and the study personnel performing post-op assessments will be blinded. Anesthesia providers cannot be blinded during this study since anesthesia providers will be required to draw up the study drugs as well as managing the wait time between rocuronium and succinylcholine. Patients are assigned to one of three groups (n = 100 each group). Each participant will undergo a standard IV induction of anesthesia (Lidocaine 1mg/kg, propofol 1-2 mg/kg titrated to effect, and succinylcholine (administered as indicated by study group assignment). Study group details are as follows: Group 1 (Control) to receive no rocuronium pretreatment and 1 mg/kg of succinylcholine. Groups 2 and 3 to receive 0.05 mg/kg up to 5 mg of rocuronium; patients ranged from 50-120 kg. In Group 2, succinylcholine administration will occur at 1.0 mg/kg at t = 1 minute after pretreatment with rocuronium. In Group 3, succinylcholine will be administered (1.0 mg/kg) at t = 2 minutes after pretreatment. The Succinylcholine-induced fasciculations will be noted on study assessment data sheet as either present or absent. . Myalgia assessment is to occur post-succinylcholine administration at t =3 hours and t = 24 hours and will be rated as described below.

Myalgia assessment:

Participants will by queried at the above time points about muscle pain and scored based on their answers as follows.

0 - no pain /no muscle stiffness

1. - mild muscle pain and/or stiffness at 1 or more sites that does not limit daily activity
2. - Moderate muscle pain and/or stiffness at 1 or more sites that does not limit daily activity
3. - Moderate generalized muscle pain and/or stiffness limiting daily activity
4. - Severe muscle pain and/or stiffness at 1 or more sites limiting movement and preventing daily activity

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective Endoscopic Retrograde Cholangiopancreatography (ERCP) under general anesthesia
* Have been informed of the nature of the study and informed consent has been obtained

Exclusion Criteria:

* Patients will be excluded if they have chronic pain requiring daily opioid use greater than 30 mg PO morphine equivalent.
* Patients will also be excluded if their comorbid medical conditions require a true rapid sequence induction as precurarization with rocuronium increases the time to intubation which is undesirable in a patient who is at high risk for aspiration.
* Patients taking muscle relaxants at home for spasticity.
* Patients under the age of 18 years old.
* Any contraindication for using succinylcholine or rocuronium.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leighan Bye, MD, Principal Investigator — Indiana University
Locations (1):
- indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martyn J, Durieux ME. Succinylcholine: new insights into mechanisms of action of an old drug. Anesthesiology. 2006 Apr;104(4):633-4. doi: 10.1097/00000542-200604000-00004. No abstract available. PMID 16571955
- [Background] Wong SF, Chung F. Succinylcholine-associated postoperative myalgia. Anaesthesia. 2000 Feb;55(2):144-52. doi: 10.1046/j.1365-2044.2000.055002144.x. PMID 10651675
- [Background] Hager HH, Burns B. Depolarizing Muscle Relaxants, Succinylcholine Chloride. [Update 2018 Jun13]. In StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2018 Jan-.
- [Background] Pace NL. Prevention of succinylcholine myalgias: a meta-analysis. Anesth Analg. 1990 May;70(5):477-83. doi: 10.1213/00000539-199005000-00002. PMID 2139549
- [Background] Motamed C, Choquette R, Donati F. Rocuronium prevents succinylcholine-induced fasciculations. Can J Anaesth. 1997 Dec;44(12):1262-8. doi: 10.1007/BF03012773. PMID 9429043
- [Background] Martin R, Carrier J, Pirlet M, Claprood Y, Tetrault JP. Rocuronium is the best non-depolarizing relaxant to prevent succinylcholine fasciculations and myalgia. Can J Anaesth. 1998 Jun;45(6):521-5. doi: 10.1007/BF03012701. PMID 9669004
- [Background] Schreiber JU, Lysakowski C, Fuchs-Buder T, Tramer MR. Prevention of succinylcholine-induced fasciculation and myalgia: a meta-analysis of randomized trials. Anesthesiology. 2005 Oct;103(4):877-84. doi: 10.1097/00000542-200510000-00027. PMID 16192781
- [Background] Abbas N, Tariq S, Khan AW, Murtaza G, Naqvi N, Khanzada A. To asses the effects of rocuronium pretreatment on succinylcholine induced fasciculations and postoperative myalgias. J Pak Med Assoc. 2009 Dec;59(12):847-50. PMID 20201179
- [Background] Kim KN, Kim KS, Choi HI, Jeong JS, Lee HJ. Optimal precurarizing dose of rocuronium to decrease fasciculation and myalgia following succinylcholine administration. Korean J Anesthesiol. 2014 Jun;66(6):451-6. doi: 10.4097/kjae.2014.66.6.451. Epub 2014 Jun 26. PMID 25006369

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Pretreated With Rocuronium: Succinylcholine administration with no Rocuronium pre-treatment
  non-pretreated Succinylcholine: no pretreatment
- Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration: Succinylcholine administration 1 minute following Rocuronium pre-treatment
  succinylcholine 1 minute after rocuronium pretreatment: 0.05 mg/kg up to 5 mg of rocuronium pretreatment followed by 1.0 mg/kg succinlycholine t = 1 min +/- 10 sec after pretreatment
- Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion: Succinylcholine administratjion 2 minutes following Rocuronium pre-treatment
  succinylcholine 2 minutes following rocuronium pretreatment: 0.05 mg/kg up to 5 mg of rocuronium pretreatment followed by 1.0 mg/kg succinlycholine t = 2 min +/- 10 sec after pretreatment.
Period: Overall Study
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Started | 100 | 100 | 100
Completed | 96 | 96 | 98
Not Completed | 4 | 4 | 2
Not completed — Protocol Violation | 4 | 3 | 2
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There is a total of 290 participants, randomized to a control arm and 2 experimental arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Not Pretreated | Pre-treated 1 Minute Before Succinylcholine Administration | Pre-treated 2 Minutes Before Succinylcholine Administratjion | Total
Number analyzed (Participants) | 96 | 96 | 98 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] — Patients age is collected upon consent as part of the demographics to be used to validate cohorts variables between arms of the study.
  years | 60 (15) | 62 (14) | 59 (16) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants] — sex/gender is collected at enrollment to use in demographic analysis between cohort groups.
  Participants
    Female | 50 | 55 | 48 | 153
    Male | 46 | 41 | 50 | 137
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Myalgias Perceived at 3 Hours
Description: The data are reported as pain (scores 1-4) vs. no pain (score 0).
Time Frame: 3 hours post succinylcholine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Number analyzed (Participants) | 96 | 96 | 98
Participants
  Patients with no pain 3 hours post succinylcholine | 81 | 83 | 83
  Patients who described having pain 3 hours post succinylcholine | 15 | 13 | 15

2. Primary Outcome: Myalgias at 24 Hours Post Succinylcholine Administration.
Description: The presence of myalgias referencing a severity scale from 0 (no muscle pain), 1 (mild muscle pain), 2(moderate muscle pain), 3 (Moderate muscle pain) and 4 (Severe muscle pain). The data are reported as pain (scores 1-4) vs. no pain (score 0)
Time Frame: 24 hours post succinylcholine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Number analyzed (Participants) | 96 | 96 | 98
Participants
  patients experiencing no pain 24 hours post succinylcholine administrations | 64 | 78 | 80
  Patients experiencing pain at 24 hours post succinylcholine administrations | 32 | 18 | 18

3. Primary Outcome: Pain Scores
Description: 0=no muscle pain/stiffness, 1=mild muscle pain/stiffness not limiting daily activity, 2=moderate muscle pain/stiffness not limiting daily activity, 3=moderate muscle pain stiffness that limits daily activity, 4=severe muscle pain/stiffness limiting movement and preventing daily activity. Values averaged.
Time Frame: 3 hours post succinylcholine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Number analyzed (Participants) | 96 | 96 | 98
Participants
  Pain score =0 | 81 | 83 | 83
  Pain score = 1 | 10 | 12 | 12
  Pain score = 2 | 4 | 1 | 2
  Pain score = 3 | 1 | 0 | 0
  Pain score = 4 | 0 | 0 | 1

4. Primary Outcome: Pain Scores
Description: as for outcome 3
Time Frame: 24 hours post succinylcholine administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Number analyzed (Participants) | 96 | 96 | 98
Participants
  24 hour pain scores = 0 | 64 | 78 | 80
  24 hour pain scores=1 | 20 | 9 | 16
  24 hour pain score=2 | 7 | 8 | 0
  24 pain score =3 | 4 | 1 | 1
  24 pain score=4 | 1 | 0 | 1

5. Secondary Outcome: Number of Participants With Observed Presence of Muscle Fasciculation Following Succinylcholine Administration
Description: Observed presence or absence of muscle fasciculation following succinylcholine administration in subjects pretreated with rocuronium 1 minute prior to succinylcholine administration or 2 minutes prior to succinylcholine administration compared to the control group not pretreated with rocuronium.
Time Frame: immediately following succinylcholine administration up to 2 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
Number analyzed (Participants) | 96 | 96 | 98
Participants | 75 | 20 | 13

ADVERSE EVENTS:
Time Frame: 24 hours post succinylcholine administration
Arm/Group | Not Pretreated With Rocuronium | Pre-treated With Rocuronium 1 Minute Before Succinylcholine Administration | Pre-treated With Rocuronium 2 Minutes Before Succinylcholine Administratjion
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT04581395/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT04581395/ICF_001.pdf